CLINICAL TRIAL: NCT03588637
Title: Real-world Effectiveness and Safety on Daptomycin in Gram-Positive Infections in Chinese Intensive Care Units
Brief Title: Real-world Daptomycin Use in Chinese ICUs
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xuelian Liao, Principal Investigator, West China Hospital
Other Study IDs: HX 00147
Record Dates: First submitted 2018-06-20; First posted 2018-07-17 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Daptomycin; Real-world Study; Intensive Care Unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patient who receive at least one dose of daptomycin
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Analyze the effectiveness and safety of Daptomycin(Jiangsu Hengrui Medicine Co., Ltd) in Gram-positive infections in Chinese Intensive Care Units by using the real-world data platform, https://rws.scccmqc.com. Patients who received at least one dose of Daptomycin between 2016 to 2021 are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received at least one dose of daptomycin

Exclusion Criteria:

* No

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are suspected of Gram-positive infection in the Intensive Care Units.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  death
Cure Rate | 30 days
  clinical and microbiological effectiveness

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 30 days
  organ dysfunction，allergy，creatine kinase levels，eosinophilic pneumonia，etc.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided